CLINICAL TRIAL: NCT02311231
Title: Bivalirudin vs Heparin in NSTEMI and STEMI in Patients on Modern Antiplatelet Therapy in SWEDEHEART A Multicenter, Prospective, Randomized Controlled Clinical Trial Based on the SWEDEHEART Platform
Brief Title: Bivalirudin vs Heparin in NSTEMI and STEMI in Patients on Modern Antiplatelet Therapy in SWEDEHEART
Acronym: VALIDATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT nr: 2012-005260-10
Record Dates: First submitted 2014-11-27; First posted 2014-12-08 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: ST-segment Elevation Myocardial Infarction; Non ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bivalirudin (Experimental): bivalirudin as intravenous bolus of 0,75 mg per kilogram followed by an infusion of 1,75 mg per kilogram per hour
  Interventions: Drug: bivalirudin
- heparin (Active Comparator): unfractionated Heparin 5 000 IU/ml as intravenous bolus according to local practice
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: bivalirudin — Will be administered as an intravenous bolus of 0.75 mg per kilogram, followed by an infusion of 1.75 mg per kilogram per hour). Bivalirudin will be administered alone or with a low dose of heparin up to 3000U heparin in lab or up to 5000 U given pre-hospital according to local practice.
  Other Names: Angiox
  Arms: bivalirudin
Drug: Heparin — Treatment with unfractionated Heparin 5000 IU/ml i.v. ,Leo Pharma, Sweden, (the control group). Heparin in the control group is administered as an intravenous or intra-arterial bolus according to local practice. A dose of 70-100 U/kg is recommended
  Other Names: Heparin 5000 IU/ml i.v. ,Leo Pharma
  Arms: heparin

SUMMARY:
In this trial we test the hypothesis that PCI and bivalirudin is superior to heparin alone (according to local protocol) in reducing death, MI, and major bleeding in patients with NSTEMI or STEMI at 180 days (primary end point), treated with ticagrelor or prasugrel.

DETAILED DESCRIPTION:
The follow up of endpoints will be performed using SWEDEHEART and national registries. Follow up of primary endpoints and stroke will also be performed by telephone contacts with the patients or first degree relatives by a nurse phone call after 7 days and 180 days. The nurses will also accumulate hospital record information on these endpoints.

A central adjudication will be performed for all reported primary endpoints for the first 180 days follow up. Every site will prepare source documents for the event and send it to UCR for central adjudication by an independent committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of NSTEMI as judged by the physician in accordance with current guideline definitions (positive troponin) or, patients with a diagnosis of STEMI as defined by chest pain suggestive for myocardial ischemia for at least 30 minutes before hospital admission, time from onset of symptoms of less than 24 hours, and an ECG with new ST-segment elevation in two or more contiguous leads of ≥0.2 mV in leads V2-V3 and/or ≥0.1 mV in other leads or a probable new-onset left bundle branch block.
* PCI of culprit lesion is intended (therapeutic PCI, not primarily diagnostic PCI).
* Treated with bolus dose of ticagrelor or prasugrel before start of PCI. See 2.6
* Ability to provide informed consent
* Age 18 years or older

Exclusion Criteria:

* Previous randomization in the VALIDATE-SWEDEHEART trial.
* Known terminal disease with life expectancy less than one year.
* Patients with known ongoing bleeding
* Patients with uncontrolled hypertension in the opinion of the investigator
* Patients with known subacute bacterial endocarditis
* Patients with known severe renal (GFR < 30 ml/min) and/or liver dysfunction
* Patients with known thrombocytopenia or thrombocyte function defects
* Any other contraindication for the study medications.
* Heparin > 5000U Before arriving to PCI lab or > 3000 U given during angiography before randomization.
* GpIIb/IIIa inhibitors have been given or are pre-planned to be given during the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6012 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Death, Myocardial infarction and major bleeding event | 180 days

SECONDARY OUTCOMES:
Death, Myocardial infarction and major bleeding events in the subgroups NSTEMI and STEMI | 180 days
Time to primary endpoints (death, myocardial infarction and major bleeding event) | 180 days
  Time to individual components of the primary end point (death, myocardial infarction and major bleeding).
Number of events where primary endpoints (death, myocardial infarction and major bleeding event) and stroke have been registered | 180 days
  The primary end point combined with stroke as reported in the Swedish national patient registry.
Number of events where primary endpoints (death, myocardial infarction and major bleeding event) have been registered in heparin subgroups (U/kg, groups with certain max ACT values etc) | 180 days
TIMI flow grade after PCI | 180 days
Time to re-hospitalization with reinfarction | 180 days
  Time to re-hospitalization with reinfarction as reported in Swedeheart
Time to all-cause death or re-hospitalization with myocardial infarction | 180 days
Time to target vessel revascularization | 180 days
  Time to target vessel revascularization as reported in SWEDEHEART.
Time to target lesion revascularization | 180 days
  Time to target lesion revascularization as reported in SWEDEHEART
Time to stent thrombosis | 180 days
  Time to stent thrombosis as reported in SWEDEHEART.
Time to restenosis | 180 days
  Time to restenosis as reported in SWEDEHEART.
Time to re-hospitalization with heart failure | 180 days
  Time to re-hospitalization with heart failure as reported in SWEDEHEART.
Heart failure and complications of PCI during index hospitalization | 180 days
  Heart failure and complications of PCI during index hospitalization as reported in SWEDEHEART
Minor bleeding during index hospitalization | 180 days
  Minor bleeding during index hospitalization as reported in SWEDEHEART
Length of index hospital stay | 180 days
  Length of index hospital stay as reported in SWEDEHEART
Bail-out use of GpIIb/IIIa | 180 days
  Bail-out use of GpIIb/IIIa inhibitors during PCI

CONTACTS AND LOCATIONS:
Overall Officials: David Erlinge, Principal Investigator — Lund University, Lund, Sweden
Locations (1):
- Lund University, Lund, Sweden

REFERENCES:
- [Derived] Omerovic E, James S, Ramundal T, Frobert O, Linder R, Danielewicz M, Hamid M, Pagonis C, Henareh L, Wagner H, Stewart J, Jensen J, Lindros P, Robertsson L, Wikstrom H, Ulvenstam A, Bhiladval P, Todt T, Ioanes D, Kellerth T, Zagozdzon L, Gotberg M, Andersson J, Angeras O, Ostlund O, Held C, Koul S, Erlinge D. Bivalirudin versus heparin in ST and non-ST-segment elevation myocardial infarction-Outcomes at two years. Cardiovasc Revasc Med. 2024 Sep;66:43-50. doi: 10.1016/j.carrev.2024.03.025. Epub 2024 Mar 26. PMID 38575449
- [Derived] James S, Koul S, Andersson J, Angeras O, Bhiladvala P, Calais F, Danielewicz M, Frobert O, Grimfjard P, Gotberg M, Henareh L, Ioanes D, Jensen J, Linder R, Lindroos P, Omerovic E, Panayi G, Ramunddal T, Sarno G, Ulvenstam A, Voltz S, Wagner H, Wikstrom H, Ostlund O, Erlinge D. Bivalirudin Versus Heparin Monotherapy in ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2021 Dec;14(12):e008969. doi: 10.1161/CIRCINTERVENTIONS.120.008969. Epub 2021 Dec 14. PMID 34903034
- [Derived] Bergman S, Mohammad MA, James SK, Angeras O, Wagner H, Jensen J, Schersten F, Frobert O, Koul S, Erlinge D. Clinical Impact of Intraprocedural Stent Thrombosis During Percutaneous Coronary Intervention in Patients Treated With Potent P2Y12 inhibitors - a VALIDATE-SWEDEHEART Substudy. J Am Heart Assoc. 2021 Sep 21;10(18):e022984. doi: 10.1161/JAHA.121.022984. Epub 2021 Sep 13. PMID 34514849
- [Derived] Rylance RT, Wagner P, Omerovic E, Held C, James S, Koul S, Erlinge D. Assessing the external validity of the VALIDATE-SWEDEHEART trial. Clin Trials. 2021 Aug;18(4):427-435. doi: 10.1177/17407745211012438. Epub 2021 May 20. PMID 34011198
- [Derived] Jamaly S, Redfors B, Omerovic E, Carlsson L, Karason K. Prognostic significance of BMI after PCI treatment in ST-elevation myocardial infarction: a cohort study from the Swedish Coronary Angiography and Angioplasty Registry. Open Heart. 2021 Feb;8(1):e001479. doi: 10.1136/openhrt-2020-001479. PMID 33589539
- [Derived] Olsson A, Ring C, Josefsson J, Eriksson A, Rylance R, Frobert O, James S, Sparv D, Erlinge D. Patient experience of the informed consent process during acute myocardial infarction: a sub-study of the VALIDATE-SWEDEHEART trial. Trials. 2020 Mar 6;21(1):246. doi: 10.1186/s13063-020-4147-0. PMID 32143733
- [Derived] Wester A, Attar R, Mohammad MA, Andell P, Hofmann R, Jensen J, Szummer K, Erlinge D, Koul S. Impact of Baseline Anemia in Patients With Acute Coronary Syndromes Undergoing Percutaneous Coronary Intervention: A Prespecified Analysis From the VALIDATE-SWEDEHEART Trial. J Am Heart Assoc. 2019 Aug 20;8(16):e012741. doi: 10.1161/JAHA.119.012741. Epub 2019 Aug 7. PMID 31387441
- [Derived] Erlinge D, Omerovic E, Frobert O, Linder R, Danielewicz M, Hamid M, Swahn E, Henareh L, Wagner H, Hardhammar P, Sjogren I, Stewart J, Grimfjard P, Jensen J, Aasa M, Robertsson L, Lindroos P, Haupt J, Wikstrom H, Ulvenstam A, Bhiladvala P, Lindvall B, Lundin A, Todt T, Ioanes D, Ramunddal T, Kellerth T, Zagozdzon L, Gotberg M, Andersson J, Angeras O, Ostlund O, Lagerqvist B, Held C, Wallentin L, Schersten F, Eriksson P, Koul S, James S. Bivalirudin versus Heparin Monotherapy in Myocardial Infarction. N Engl J Med. 2017 Sep 21;377(12):1132-1142. doi: 10.1056/NEJMoa1706443. Epub 2017 Aug 27. PMID 28844201